CLINICAL TRIAL: NCT06407960
Title: The Clinical Study of the Reliability and Validity of the Foot Function Index in the Application of Pediatric and Adolescent Flatfoot, and Its Correlation With Dynamic Plantar Pressure
Brief Title: The Clinical Study of Foot Function Index in Adolescent Flatfoot
Status: Completed | Type: Observational
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2022-T125-2
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-01

CONDITIONS: Foot Function Index, Flat Foot, Dynamic Plantar Pressure, Reliability, Validity
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Using dynamic plantar pressure data during walking, combined with the FFI scores of adolescents, aids doctors and rehabilitation therapists in conducting more accurate, objective, and scientific evaluations of the functional parameters of the foot for appropriate rehabilitation treatment. Clinical studies on flat feet mainly focus on imaging diagnosis, gait characteristics, orthopedic insole studies, and different surgical treatment schemes related to flat foot injuries. However, few studies have analyzed the dynamic plantar pressure characteristics of flat feet to guide clinical interventions, as well as the correlation between the subjective perception of FFI and objective biomechanical parameter characteristics to analyze the validity of FFI and elucidate the physiological characteristics of foot diseases.

Specific purpose of this study Therefore, the purpose of our study was to clarify the reliability and validity of the application of the FFI in flatfoot and the correlation between the FFI and dynamic plantar pressure.

ELIGIBILITY:
Inclusion Criteria:

7-18 years old. Arch development begins to stabilize around age 7 [19]; therefore, preschool children under 7 were excluded. Ability to maintain a static standing posture unassisted; bilateral flexible flatfoot (where the heel is valgus and the arch collapses on both sides); no congenital malformation or injury of the lower limbs; normal body mass index (BMI); no previous surgery or corrective treatment for flatfoot problems; and no obvious abnormal gait and posture.

Exclusion Criteria:

Preschool children under 7 years of age are excluded. ① Foot fracture or surgical history in the past six months; ② There are muscular nervous system diseases and syndrome affecting gait and posture, such as knee valgus, knee varus, legs unequal length or scoliosis; ③BMI≥28 kg/m².

Ages: 7 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Ninety-seven participants were enrolled in this study: 41 in the flatfoot observation group and 56 in the healthy control group. The mean age of all participants was 12.990±3.187 years, height 155.976±22.649 cm, weight 52.299±15.888 kg, BMI 20.5±3.405 kg/m2, and the percentage of male participants was 41.237%.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The FFI questionnaire | The first week
  The FFI comprises 23 questions divided into 3 subdomains to evaluate the impact of foot pathology: pain (9 questions), disability (9 questions), and activity restrictions (5 questions). In combination with the visual analog scale, each question was assigned a score of 0-10 (0 for no pain or difficulty and 10 for maximum pain or difficulty).

SECONDARY OUTCOMES:
Plantar stress test | The first week
  Plantar pressure data were detected and acquired exclusively from the patients. The main outcome measures included contact area, peak pressure, and peak force.

OTHER OUTCOMES:
Physical consultation | The first week
  we measured radiography images of the Meary and pitch angles using the picture archiving and communication system (PACS) of the hospital imaging platform to determine flatfoot severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Traditional Chinese Medicine, Shanghai, Shanhai, China